CLINICAL TRIAL: NCT05373615
Title: Effect of Continuous Renal Replacement Therapy and Residual Renal Clearance on Cefiderocol Pharmacokinetics in Critically Ill Adult Patients
Brief Title: Cefiderocol Plasma Concentrations in Patients Receiving Renal Replacement Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Shionogi Inc. (Industry)
Responsible Party: Principal Investigator, Tomefa Asempa, Associate Director, Clinical and Translational Infectious Diseases Research, Hartford Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HHC-2022-0045
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Cefiderocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cefiderocol (Experimental): Participants will receive four to six doses of Cefiderocol as per current prescribing information based on effluent rate
  Interventions: Drug: Cefiderocol

INTERVENTIONS:
Drug: Cefiderocol — After receipt of Cefiderocol, blood samples will be collected at various time points to determine the pharmacokinetics of Cefiderocol

SUMMARY:
Continuous renal replacement therapies (CRRT) such as continuous venovenous hemofiltration are used to provide renal support for critically ill patients with acute kidney injury (AKI), particularly patients who are hemodynamically unstable. It is well known that critically ill patients may experience alterations in antibiotic pharmacokinetics, and as a result, dosing modifications are generally required. There is a need to understand how CRRT affect the pharmacokinetics and disposition of drugs. This study is designed to assess the pharmacokinetics of the new broad-spectrum antibiotic, Cefiderocol, in critically ill patient receiving CRRT.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, Phase 1b, pharmacokinetic study of Cefiderocol in 16 critically ill patients receiving CRRT support. Informed consent will be collected from all study participants, legal authorized representative, or their next of kin in order to participate. This is not a treatment study; all participants will receive standard of care antibiotics which may include cefiderocol as necessary to treat any current infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Receiving CRRT including CVVH, CVVHD, and CVVHDF support.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding;
2. History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic (a history of mild rash to a cephalosporin followed by uneventful re-exposure is not a contraindication);
3. A hemoglobin less than 8 gm/dl at baseline;
4. Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal;
5. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator);
6. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Cefiderocol concentration | 8 to 12 hours
  The total and free plasma concentration of cefiderocol over time
Cefiderocol clearance | 8 to 12 hours
  The Clearance in liters/hour of Cefiderocol from the plasma
Cefiderocol maximum concentration | 8 to 12 hours
  The maximum concentration of Cefiderocol from the plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No